CLINICAL TRIAL: NCT06485323
Title: MRI Pseudo-CT Sequences for Obstetrical Pelvimetry
Acronym: Pelvi-MRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023/07AVR/174
Record Dates: First submitted 2024-05-27; First posted 2024-07-03 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Obstetric Labor Complications
Keywords: technological progress
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Intervention Model Description: Each patients will have a CT scan (classic follow-up) and an MRI (for the study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IRM + CT scan for Pelvimetry (Experimental)
  Interventions: Device: MRI pelvimetry

INTERVENTIONS:
Device: MRI pelvimetry — MRI of the pelvis

SUMMARY:
It is possible to perform a pelvimetry by MRI as a substitute to pelvimetry by CT, hence sparing the patient from a dose of irradiation.

DETAILED DESCRIPTION:
The Principal investigator want to evaluate new MRI sequences offering both an optimal contrast between mineral bone and soft tissues, and a shorter acquisition time. Indeed, the recent developments of specific MRI sequences to preferentially image the mineral bone (namely the ZTE and lavaflex 3D T1-weighted SPGR sequences) allow performing pelvimetry measurements on MR images offering an optimal "pseudo CT" contrast, with an MR acquisition time that is less than 10 minutes. Preliminary tests of these sequences have been carried out in our center in order to be able to implement these sequences on our clinical and research MRI machines. The study team wish to undertake a study to validate the use of this rapid and non-irradiating MRI approach, with the aim to replace a CT pelvimetry by a MRI pelvimetry demonstrated as being as reliable.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman 33 to 41 week
* Woman who gave birth by cesarean section, for whom the obstetrician requests a pelvimetry CT for the next pregnancy
* Pelvimetry planned by the obstetrical team outside of "emergency" pathway
* Adhere to the study protocol after reading the patient information document have signed the informed consent form to participate in the study

Exclusion Criteria:

* Usual contraindications to MRI (Pacemaker, Metallic foreign body, Cochlear implant,…)
* Severe claustrophobia
* uncomfortable back position

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — having an uterus
Enrollment: 95 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prove the non-inferiority of MRI compared to CT for pelvimetry. | 30 minutes (duration of the exam+ measurement)
  Measurement of pelvic bone diameters in pregnant women

SECONDARY OUTCOMES:
Evaluate patient convenience for both examinations (CT and MRI) | immediately after both examinations
  questionnaire (scale from zero to ten, zero = more pleasant, ten=least pleasant)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Lecouvet, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universaires Siant Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hampel F, Hallscheidt P, Sohn C, Schlehe B, Brocker KA. Pelvimetry in nulliparous and primiparous women using 3 Tesla magnetic resonance imaging. Neurourol Urodyn. 2018 Aug;37(6):1950-1956. doi: 10.1002/nau.23537. Epub 2018 Feb 21. PMID 29464757
- [Background] Li J, Lou Y, Chen C, Zheng W, Chen Y, Dong T, Yang M, Zhao B, Luo Q. Predictive Value of MRI Pelvimetry in Vaginal Delivery and Its Practicability in Prolonged Labour-A Prospective Cohort Study. J Clin Med. 2023 Jan 5;12(2):442. doi: 10.3390/jcm12020442. PMID 36675370
- [Background] Liao KD, Yu YH, Li YG, Chen L, Peng C, Liu P, Chen CL, Chen RY, Zhong M, Wang Y. Three-dimensional magnetic resonance pelvimetry: A new technique for evaluating the female pelvis in pregnancy. Eur J Radiol. 2018 May;102:208-212. doi: 10.1016/j.ejrad.2018.03.024. Epub 2018 Mar 19. PMID 29685537